CLINICAL TRIAL: NCT05758350
Title: Effect of Home Based Swallowing Exercise in Stroke Patients With Dysphagia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CF22483A
Record Dates: First submitted 2023-02-21; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Dysphagia Following Cerebrovascular Accident
Keywords: dysphagia; ischemic stroke; intracranial hemorrhage
MeSH Terms: conditions — Deglutition Disorders; Ischemic Stroke; Intracranial Hemorrhages

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iowa Oral Performance Instrument (IOPI) training group (Experimental): Including conventional speech therapy (tongue range of motion and strength, oral diet suggestion, masseter muscle strengthening) and home- IOPI based resistance training
  Interventions: Behavioral: home based IOPI swallow training
- controlled group (No Intervention): Including conventional speech therapy (tongue range of motion and strength, oral diet suggestion, masseter muscle strengthening) only

INTERVENTIONS:
Behavioral: home based IOPI swallow training — Use IOPI for tongue and labial muscle resistance training. Conventional training was the same as controlled group.
  Arms: Iowa Oral Performance Instrument (IOPI) training group

SUMMARY:
Dysphagia is a common problem in post-stroke patients and greatly impaired quality of life. Among them, the strength of tongue and lip muscles played a key role in the oral phase of swallowing and many stroke survivors suffered from these muscles weakness. Iowa oral performance instrument (IOPI) is a standardized portable device that can be used to quantify tongue muscle strength, thus allowing the clinician to set the level of resistance necessary to achieve optimal gains in strength, and also providing visual feedback of performance to the patients to guide training. In this study, we use Videofluoroscopic Swallowing Study (VFSS) to screen for the stroke patient suffering from dysphagia and recruited them into the trial. They then participated in a home based resistance-training program using the tongue depressor, 1 time everyday and each time consisted of 30 repetitions, totally 4 weeks. Various tongue strength variables and subjective scale were obtained before and after the intervention. The purpose of the study was to evaluate the effect of the home based swallowing therapy in the post stroke dysphagia patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke within 1 year, videofluoroscopic swallow study revealed abnormalities
* Mini-Mental Status Examination >20, could cooperate swallow therapy

Exclusion Criteria:

* Already known dysphagia before stroke event
* Malocclusion or severe facial palsy
* Localized oral lesion interfering swallowing

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Anterior tongue pressure | 1 week after treatment
Posterior tongue pressure | 1 week after treatment
Right buccal pressure | 1 week after treatment
Left buccal pressure | 1 week after treatment
Labial pressure | 1 week after treatment

SECONDARY OUTCOMES:
The score of Eat-10 scale | 1 week after treatment

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee JH, Kim HS, Yun DH, Chon J, Han YJ, Yoo SD, Kim DH, Lee SA, Joo HI, Park JS, Kim JC, Soh Y. The Relationship Between Tongue Pressure and Oral Dysphagia in Stroke Patients. Ann Rehabil Med. 2016 Aug;40(4):620-8. doi: 10.5535/arm.2016.40.4.620. Epub 2016 Aug 24. PMID 27606268
- [Background] Park JS, Kim HJ, Oh DH. Effect of tongue strength training using the Iowa Oral Performance Instrument in stroke patients with dysphagia. J Phys Ther Sci. 2015 Dec;27(12):3631-4. doi: 10.1589/jpts.27.3631. Epub 2015 Dec 28. PMID 26834320
- [Background] Park HS, Oh DH, Yoon T, Park JS. Effect of effortful swallowing training on tongue strength and oropharyngeal swallowing function in stroke patients with dysphagia: a double-blind, randomized controlled trial. Int J Lang Commun Disord. 2019 May;54(3):479-484. doi: 10.1111/1460-6984.12453. Epub 2019 Jan 28. PMID 30693627
- [Result] Kim HD, Choi JB, Yoo SJ, Chang MY, Lee SW, Park JS. Tongue-to-palate resistance training improves tongue strength and oropharyngeal swallowing function in subacute stroke survivors with dysphagia. J Oral Rehabil. 2017 Jan;44(1):59-64. doi: 10.1111/joor.12461. PMID 27883209